CLINICAL TRIAL: NCT05064358
Title: A Phase 2, Randomized, Parallel, Open-label Study to Investigate the Safety, Efficacy, and Pharmacokinetics of Various Dosing Regimens of Single-agent Belantamab Mafodotin (GSK2857916) in Participants With Relapsed or Refractory Multiple Myeloma (DREAMM-14)
Brief Title: Study to Investigate Alternative Dosing Regimens of Belantamab Mafodotin in Participants With Relapsed or Refractory Multiple Myeloma
Acronym: DREAMM 14
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 209628; 2021-004151-16 (EudraCT Number); 2023-508213-16 (Registry Identifier: CTIS)
Record Dates: First submitted 2021-09-22; First posted 2021-10-01 (Actual); Results first posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Multiple Myeloma
Keywords: Antibody drug conjugate; Belantamab mafodotin; BLENREP; DREAMM14; GSK2857916; Alternative dosing; Relapsed or refractory multiple myeloma; RRMM
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — belantamab mafodotin

STUDY DESIGN:
Intervention Model Description: Belantamab mafodotin will be administered using various dosing regimens.
Masking Description: It is an open label study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1: Participants receiving belantamab mafodotin at dose level (DL) 1 (Experimental)
  Interventions: Drug: Belantamab mafodotin
- Cohort 2: Participants receiving belantamab mafodotin at DL 2 (Experimental)
  Interventions: Drug: Belantamab mafodotin
- Cohort 3: Participants receiving belantamab mafodotin at DL 3 (Experimental)
  Interventions: Drug: Belantamab mafodotin
- Cohort 4: Participants receiving belantamab mafodotin at DL 4 (Experimental)
  Interventions: Drug: Belantamab mafodotin
- Cohort 5: Participants receiving belantamab mafodotin at DL4 with alternative dose modification (Experimental)
  Interventions: Drug: Belantamab mafodotin

INTERVENTIONS:
Drug: Belantamab mafodotin — Belantamab mafodotin will be administered.

SUMMARY:
This study aims to evaluate alternative dosing regimens of single-agent belantamab mafodotin in participants with relapsed or refractory multiple myeloma (RRMM) to determine if an improved overall benefit/risk profile can be achieved by modifying the belantamab mafodotin dose, schedule, or both.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 years of age inclusive at the time of signing the informed consent form (ICF).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
* Histologically or cytologically confirmed diagnosis of MM and a. Has undergone stem cell transplant or is considered transplant ineligible, and b. Has failed at least 3 prior lines of anti-myeloma therapies, including an anti-cluster of differentiation (CD)38 antibody (e.g., daratumumab) alone or in combination and is refractory to an immunomodulatory agent (e.g., lenalidomide, pomalidomide) and a proteasome inhibitor (e.g., bortezomib, ixazomib, carfilzomib).
* France specific: participants have failed at least 4 prior lines of anti-myeloma therapies
* Participant has measurable disease per modified IMWG criteria.
* Life expectancy of at least 6 months, in the opinion of the investigator.
* Male and female participants agree to abide by protocol-defined contraceptive requirements.
* Participant is capable of giving signed informed consent.
* Participant meets country-specific inclusion criteria described in the protocol.

Exclusion Criteria:

* Symptomatic amyloidosis, active POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, myeloma protein, and skin changes), or active plasma cell leukemia at the time of screening.
* Current corneal epithelial disease, except nonconfluent superficial punctate keratitis (SPK).
* Evidence of active mucosal or internal bleeding.
* Presence of an active renal condition.
* Any serious and/or unstable pre-existing medical condition, psychiatric disorder, or other conditions that could interfere with the participant's safety, obtaining informed consent, or compliance with the study procedures.
* Malignancies other than the disease under study, except for any other malignancy from which the participant has been disease free for >2 years and, will not affect the evaluation of the effects of the study treatment on the currently targeted malignancy (MM). Participants with curatively treated non-melanoma skin cancer may be enrolled without a 2-year restriction.
* Evidence of cardiovascular risk as per the protocol criteria.
* Pregnant or lactating female.
* Active infection requiring antibiotic, antiviral, or antifungal treatment.
* Known human immunodeficiency virus (HIV) infection, unless the criteria in protocol can be met.
* Hepatitis B and C will be excluded unless the criteria in protocol can be met.
* Cirrhosis or current unstable liver or biliary disease.
* Alanine aminotransferase (ALT) >2.5× upper limit of normal (ULN).
* Total Bilirubin >1.5×ULN.
* Systemic anti-MM therapy within <=14 days or 5 half-lives, whichever is shorter.
* Systemic therapy with high dose steroids within <=14 days before the first dose of study treatment.
* Prior allogenic stem cell transplant.
* Prior treatment with a monoclonal antibody <=30 days before the first dose of study treatment. Use of monoclonal antibodies for serious conditions unrelated to multiple myeloma, such as COVID, may be permitted.
* Prior treatment with an anti-B cell maturation antigen (BCMA) targeted therapy or hypersensitivity reactions to any components of the study treatment.
* Treatment with an antibody-drug conjugate.
* Participant has received any major surgery <=4 weeks before the first dose of study treatment. An exception may be allowed for bone stabilizing surgery.
* Inadequate bone marrow reserve or organ functions as demonstrated by any of the following: a. Absolute neutrophil count <1.0×10^9/L, b. Hemoglobin <8 gram/deciliter (g/dL), c. Platelet count <50×10^9/L, d. Spot urine (albumin/creatinine ratio) >500 milligram/gram (mg/g), e. Estimated glomerular filtration rate (eGFR) <30 milliliter per minute per 1.73 meter square (mL/min/1.73m^2).
* UK specific: a. Absolute neutrophil count <1.5×10^9/L, c. Platelet count <75×10^9/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2024-08-19 (Actual); Study Completion 2026-01-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (78):
- United States (6):
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Chattanooga, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Houston, Texas
- Argentina (5):
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Capital Federal
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aire
  - GSK Investigational Site, Pilar
  - GSK Investigational Site, Rosario
- Australia (4):
  - GSK Investigational Site, Liverpool, New South Wales
  - GSK Investigational Site, Newcastle, New South Wales
  - GSK Investigational Site, Woodville, South Australia
  - GSK Investigational Site, East Melbourne, Victoria
- Brazil (5):
  - GSK Investigational Site, Joinville
  - GSK Investigational Site, Porto Alegre
  - GSK Investigational Site, Rio de Janeiro
  - GSK Investigational Site, Salvador
  - GSK Investigational Site, São Paulo
- Canada (3):
  - GSK Investigational Site, Oshawa, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
- France (3):
  - GSK Investigational Site, Avignon
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Orléans
- Germany (4):
  - GSK Investigational Site, Cottbus
  - GSK Investigational Site, Dresden
  - GSK Investigational Site, Greifswald
  - GSK Investigational Site, Hamburg
- Greece (2):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Rio Patras
- India (7):
  - GSK Investigational Site, Ahmedabad
  - GSK Investigational Site, Apex Wellness Hospital
  - GSK Investigational Site, Hyderabad
  - GSK Investigational Site, Kolkata
  - GSK Investigational Site, M S R Nagar Msrit Post
  - GSK Investigational Site, Pune
  - GSK Investigational Site, Sushrut Hospital and Research
- GSK Investigational Site, Dublin, Ireland
- Italy (8):
  - GSK Investigational Site, Alessandria
  - GSK Investigational Site, Ascoli Piceno
  - GSK Investigational Site, Cagliari
  - GSK Investigational Site, Ferrara
  - GSK Investigational Site, Genova
  - GSK Investigational Site, Meldola FC
  - GSK Investigational Site, Reggio Emilia
  - GSK Investigational Site, Rimini
- GSK Investigational Site, Mexico City, Mexico
- Poland (9):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Katowice
  - GSK Investigational Site, Lublin
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Torun
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Wałbrzych
  - GSK Investigational Site, Wroclaw
- South Korea (3):
  - GSK Investigational Site, Hwasun
  - GSK Investigational Site, Pusan
  - GSK Investigational Site, Seoul
- Spain (7):
  - GSK Investigational Site, Albacete
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Girona
  - GSK Investigational Site, Oviedo
  - GSK Investigational Site, Terrassa - Barcelona
  - GSK Investigational Site, Valencia
- GSK Investigational Site, Bern, Switzerland
- Taiwan (3):
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Tainan
  - GSK Investigational Site, Taipei
- Thailand (3):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Chiang Mai
  - GSK Investigational Site, Khon Kaen
- United Kingdom (3):
  - GSK Investigational Site, Leicester
  - GSK Investigational Site, London
  - GSK Investigational Site, Stoke-on-Trent

IPD SHARING:
Plan to Share IPD: No
GSK will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The results presented are based on the data cut-off date of 30 Jan 2025. Those participants still benefiting from study drug in the opinion of their treating physician continued to receive study drug in the Post Analysis Continuation of Treatment (PACT) phase. Additional safety results will be provided within one year of study completion.
Groups:
- Arm A: Belantamab Mafodotin 2.5 Milligram (mg)/Kilogram (kg) Every 3 Weeks (Q3W): Participants with Relapsed or Refractory Multiple Myeloma (RRMM) received belantamab mafodotin as 2.5 milligram (mg)/kilogram (kg) dose on Day 1 of every 3 weeks (Q3W) as a 30-60 minute intravenous (IV) infusion until confirmed disease progression, unacceptable toxicity or death.
- Arm B: Belantamab Mafodotin 1.9 mg/kg Q3W: Participants with RRMM received belantamab mafodotin as 1.9 mg/kg dose on Day 1 of Q3W as a 30-60 minute IV infusion until confirmed disease progression, unacceptable toxicity or death.
- Arm C: Belantamab Mafodotin 2.5 mg/kg Every 6 Weeks (Q6W): Participants with RRMM received belantamab mafodotin as 2.5 mg/kg dose on Day 1 of every 6 weeks (Q6W) as a 30-60 minute IV infusion until confirmed disease progression, unacceptable toxicity or death.
- Arm D: Belantamab Mafodotin 1.9 mg/kg Q6W: Participants with RRMM received belantamab mafodotin as 1.9 mg/kg dose on Day 1 of Q6W as a 30-60 minute IV infusion until confirmed disease progression, unacceptable toxicity or death.
- Arm E: Belantamab Mafodotin 1.9 mg/kg Q6W (Based on OSDI + Visual Acuity [VA] Assessment): Participants with RRMM received belantamab mafodotin as 1.9 mg/kg dose on Day 1 of Q6W as a 30-60 minute IV infusion until confirmed disease progression, unacceptable toxicity or death. For this arm, dose modification decisions were determined by the results of the Ocular Surface Disease Index (OSDI) questionnaire or VA assessments using Snellen chart. The OSDI scale assesses the severity of eye symptoms and their impact and Snellen chart is for the assessment of visual acuity.
Period: Overall Study
Arm/Group | Arm A: Belantamab Mafodotin 2.5 Milligram (mg)/Kilogram (kg) Every 3 Weeks (Q3W) | Arm B: Belantamab Mafodotin 1.9 mg/kg Q3W | Arm C: Belantamab Mafodotin 2.5 mg/kg Every 6 Weeks (Q6W) | Arm D: Belantamab Mafodotin 1.9 mg/kg Q6W | Arm E: Belantamab Mafodotin 1.9 mg/kg Q6W (Based on OSDI + Visual Acuity [VA] Assessment)
Started (Intent-to-Treat Population included all randomized participants, whether or not randomized treatment was administered.) | 40 | 40 | 40 | 40 | 17
Safety (All randomized participants who received at least 1 dose of study treatment.) | 39 | 40 | 39 | 40 | 17
Pharmacokinetic (All participants in the Safety Population from whom at least 1 post-treatment pharmacokinetic (PK) sample was obtained and analyzed.) | 38 | 41 (1 participant was randomized in Arm A but inadvertently given Arm B treatment at Cycle 1.) | 39 | 40 | 17
Completed | 10 | 7 | 8 | 9 | 7
Not Completed | 30 | 33 | 32 | 31 | 10
Not completed — Death | 23 | 23 | 25 | 21 | 5
Not completed — Lost to Follow-up | 1 | 2 | 0 | 2 | 0
Not completed — Physician Decision | 1 | 1 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 5 | 3 | 6 | 3
Not completed — Ongoing at the time of analysis | 1 | 2 | 2 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Belantamab Mafodotin 2.5 Milligram (mg)/Kilogram (kg) Every 3 Weeks (Q3W) | Arm B: Belantamab Mafodotin 1.9 mg/kg Q3W | Arm C: Belantamab Mafodotin 2.5 mg/kg Every 6 Weeks (Q6W) | Arm D: Belantamab Mafodotin 1.9 mg/kg Q6W | Arm E: Belantamab Mafodotin 1.9 mg/kg Q6W (Based on OSDI + Visual Acuity [VA] Assessment) | Total
Number analyzed (Participants) | 40 | 40 | 40 | 40 | 17 | 177
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 66.6 (10.36) | 63.0 (9.02) | 63.7 (9.92) | 65.4 (8.87) | 67.1 (10.42) | 64.9 (9.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 21 | 19 | 16 | 8 | 83
  Male | 21 | 19 | 21 | 24 | 9 | 94
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 9 | 12 | 6 | 6 | 46
  Not Hispanic or Latino | 27 | 31 | 28 | 34 | 11 | 131

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Grade ≥2 Corneal Events Assessed by Keratopathy Visual Acuity (KVA) Scale
Description: The KVA scale is based on the evaluation of corneal changes using slit lamp examination. This scale provides a standardized approach for evaluating the relationship between corneal health and visual acuity. KVA scale is defined as Grade 0: No keratopathy, normal visual acuity with no corneal abnormalities; Grade 1: Mild changes to the cornea with no significant loss in visual acuity; Grade 2: Moderate corneal changes with noticeable visual acuity reduction; Grade 3: Severe corneal changes with substantial visual acuity impairment; Grade 4: Very severe corneal changes leading to significant vision loss. Higher grade indicates greater severity of corneal events.
Time Frame: Up to 29.5 months
Population: Safety Population included all randomized participants who received at least 1 dose of study treatment. As outlined in the protocol, the objective was to examine the corneal events in Arms B to D, compared to Arm A; hence, Arm E was not included.
Measure: Number; unit: Percentage of participants
Arm/Group | Arm A: Belantamab Mafodotin 2.5 Milligram (mg)/Kilogram (kg) Every 3 Weeks (Q3W) | Arm B: Belantamab Mafodotin 1.9 mg/kg Q3W | Arm C: Belantamab Mafodotin 2.5 mg/kg Every 6 Weeks (Q6W) | Arm D: Belantamab Mafodotin 1.9 mg/kg Q6W
Number analyzed (Participants) | 39 | 40 | 39 | 40
Percentage of participants | 64 | 40 | 44 | 38

2. Secondary Outcome: Number of Participants With Corneal Events up to Week 16
Description: The number of participants with corneal events were assessed using KVA scale. The KVA scale provides a standardized approach for evaluating the relationship between corneal health and visual acuity. KVA scale is defined as Grade 0: No keratopathy, normal visual acuity with no corneal abnormalities; Grade 1: Mild changes to the cornea with no significant loss in visual acuity; Grade 2: Moderate corneal changes with noticeable visual acuity reduction; Grade 3: Severe corneal changes with substantial visual acuity impairment; Grade 4: Very severe corneal changes leading to significant vision loss. Higher grade indicates greater severity of corneal events.
Time Frame: Up to week 16
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Belantamab Mafodotin 2.5 Milligram (mg)/Kilogram (kg) Every 3 Weeks (Q3W) | Arm B: Belantamab Mafodotin 1.9 mg/kg Q3W | Arm C: Belantamab Mafodotin 2.5 mg/kg Every 6 Weeks (Q6W) | Arm D: Belantamab Mafodotin 1.9 mg/kg Q6W | Arm E: Belantamab Mafodotin 1.9 mg/kg Q6W (Based on OSDI + Visual Acuity [VA] Assessment)
Number analyzed (Participants) | 39 | 40 | 39 | 40 | 17
Participants | 26 | 25 | 23 | 24 | 12

3. Secondary Outcome: Incidence Rate of Corneal Events by Grade (KVA Scale)
Description: Incidence rate of corneal events is defined as the percentage of participants with corneal events by grade according to the KVA scale. The KVA scale provides a standardized approach for evaluating the relationship between corneal health and visual acuity. KVA scale is defined as Grade 0: No keratopathy, normal visual acuity with no corneal abnormalities; Grade 1: Mild changes to the cornea with no significant loss in visual acuity; Grade 2: Moderate corneal changes with noticeable visual acuity reduction; Grade 3: Severe corneal changes with substantial visual acuity impairment; Grade 4: Very severe corneal changes leading to significant vision loss. Higher grade indicates greater severity of corneal events.
Time Frame: Up to 152 weeks
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Arm A: Belantamab Mafodotin 2.5 Milligram (mg)/Kilogram (kg) Every 3 Weeks (Q3W) | Arm B: Belantamab Mafodotin 1.9 mg/kg Q3W | Arm C: Belantamab Mafodotin 2.5 mg/kg Every 6 Weeks (Q6W) | Arm D: Belantamab Mafodotin 1.9 mg/kg Q6W | Arm E: Belantamab Mafodotin 1.9 mg/kg Q6W (Based on OSDI + Visual Acuity [VA] Assessment)
Number analyzed (Participants) | 39 | 40 | 39 | 40 | 12
Percentage of participants
  Grade 1 | 3 | 10 | 7 | 10 | 2
  Grade 2 | 10 | 4 | 5 | 6 | 3
  Grade 3 | 15 | 9 | 11 | 9 | 6
  Grade 4 | 0 | 3 | 1 | 0 | 2

4. Secondary Outcome: Exposure Adjusted Incidence Rate of Corneal Events as Per CTCAE Grade
Description: Exposure adjusted incidence rate of corneal events is defined as the number of participants with corneal events divided by the total exposure time for all participants at risk in the treatment group. Incidence rate for corneal events was assessed using Common Terminology Criteria for Adverse Events (CTCAE). Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe or medically significant but not immediately life-threatening; Grade 4: Life-threatening consequences; Grade 5: Death related to AE. Higher grades indicate greater severity. The number of participants with Grades 3,4, and 5 are presented.
Time Frame: Up to 152 weeks
Population: Safety Population
Measure: Number; unit: Events per 100 patient years
Arm/Group | Arm A: Belantamab Mafodotin 2.5 Milligram (mg)/Kilogram (kg) Every 3 Weeks (Q3W) | Arm B: Belantamab Mafodotin 1.9 mg/kg Q3W | Arm C: Belantamab Mafodotin 2.5 mg/kg Every 6 Weeks (Q6W) | Arm D: Belantamab Mafodotin 1.9 mg/kg Q6W | Arm E: Belantamab Mafodotin 1.9 mg/kg Q6W (Based on OSDI + Visual Acuity [VA] Assessment)
Number analyzed (Participants) | 39 | 40 | 39 | 40 | 17
Events per 100 patient years
  Grade 3 | 4 | 2 | 4 | 0 | 3
  Grade 4 | 0 | 0 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Median Duration of All the Dose Delays
Description: Median duration of dose delays is defined as the median duration in time of all the dose delays in the respective treatment group. Duration of delays is defined as period from the expected start date of dose to actual start date of current dose.
Time Frame: Up to 152 weeks
Population: Safety Population
Measure: Median (Full Range); unit: Days
Arm/Group | Arm A: Belantamab Mafodotin 2.5 Milligram (mg)/Kilogram (kg) Every 3 Weeks (Q3W) | Arm B: Belantamab Mafodotin 1.9 mg/kg Q3W | Arm C: Belantamab Mafodotin 2.5 mg/kg Every 6 Weeks (Q6W) | Arm D: Belantamab Mafodotin 1.9 mg/kg Q6W | Arm E: Belantamab Mafodotin 1.9 mg/kg Q6W (Based on OSDI + Visual Acuity [VA] Assessment)
Number analyzed (Participants) | 39 | 40 | 39 | 40 | 17
Days | 39.0 [16 to 144] | 18.0 [4 to 125] | 51.0 [18 to 163] | 60.0 [34 to 103] | 59.0 [25 to 88]

6. Secondary Outcome: Percentage of Participants Requiring Dose Reduction, Dose Interruption/Delay, Permanent Treatment Discontinuation Due to Corneal Events
Description: The percentage of participants that required dose reduction, dose interruption/delay, permanent treatment discontinuation due to corneal events were evaluated using KVA Scale. KVA scale is defined as Grade 0: No keratopathy, normal visual acuity with no corneal abnormalities; Grade 1: Mild changes to the cornea with no significant loss in visual acuity; Grade 2: Moderate corneal changes with noticeable visual acuity reduction; Grade 3: Severe corneal changes with substantial visual acuity impairment; Grade 4: Very severe corneal changes leading to significant vision loss. Higher grade indicates greater severity of corneal events.
Time Frame: Up to 152 weeks
Population: Safety Population. Only those participants who experienced corneal events have been analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Arm A: Belantamab Mafodotin 2.5 Milligram (mg)/Kilogram (kg) Every 3 Weeks (Q3W) | Arm B: Belantamab Mafodotin 1.9 mg/kg Q3W | Arm C: Belantamab Mafodotin 2.5 mg/kg Every 6 Weeks (Q6W) | Arm D: Belantamab Mafodotin 1.9 mg/kg Q6W | Arm E: Belantamab Mafodotin 1.9 mg/kg Q6W (Based on OSDI + Visual Acuity [VA] Assessment)
Number analyzed (Participants) | 26 | 25 | 23 | 24 | 12
Percentage of participants
  Dose Reduction | 31 | 28 | 26 | 23 | 35
  Dose Interruption/Delay | 59 | 35 | 28 | 33 | 29
  Permanent Treatment Discontinuation | 0 | 3 | 0 | 0 | 6

7. Secondary Outcome: Cumulative Incidence of Grade 2 or Above Corneal Events (KVA Scale)
Description: Cumulative incidence of Grade 2 or above corneal events is defined as the percentage of corneal events of Grade 2 or above, as assessed using the KVA scale, within a specific time interval. KVA scale is defined as Grade 0: No keratopathy, normal visual acuity with no corneal abnormalities; Grade 1: Mild changes to the cornea with no significant loss in visual acuity; Grade 2: Moderate corneal changes with noticeable visual acuity reduction; Grade 3: Severe corneal changes with substantial visual acuity impairment; Grade 4: Very severe corneal changes leading to significant vision loss. Higher grade indicates greater severity of corneal events.
Time Frame: At 3 months, 6 months, 9 months and 12 months
Population: Safety Population. Only those participants who experienced corneal events (KVA scale) of Grade 2 or above have been analyzed.
Measure: Number; unit: Percentage of events
Arm/Group | Arm A: Belantamab Mafodotin 2.5 Milligram (mg)/Kilogram (kg) Every 3 Weeks (Q3W) | Arm B: Belantamab Mafodotin 1.9 mg/kg Q3W | Arm C: Belantamab Mafodotin 2.5 mg/kg Every 6 Weeks (Q6W) | Arm D: Belantamab Mafodotin 1.9 mg/kg Q6W | Arm E: Belantamab Mafodotin 1.9 mg/kg Q6W (Based on OSDI + Visual Acuity [VA] Assessment)
Number analyzed (Participants) | 25 | 16 | 17 | 15 | 11
Percentage of events
  At 3 months | 59 | 32 | 36 | 33 | 53
  At 6 months | 64 | 37 | 41 | 38 | 59
  At 9 months | 64 | 40 | 41 | 38 | 59
  At 12 months | 64 | 40 | 44 | 38 | 59

8. Secondary Outcome: Toxicity Index (TI)
Description: Toxicity Index is a composite score derived from the severity grades of adverse events (AEs) reported during the study, based on the Common Terminology Criteria for Adverse Events (CTCAE). A participant's score is calculated as a function of the ordered toxicity grades, represented in descending order by sequence, on a scale of 0-6, where 0 represents no toxicity and 6 represents the highest toxicity. CTCAE grades are defined as follows: Grade 1 (Mild), Grade 2 (Moderate), Grade 3 (Severe or medically significant but not immediately life-threatening), Grade 4 (Life-threatening consequences), and Grade 5 (Death related to AE). Higher grades indicate greater toxicity severity.
Time Frame: Up to 152 weeks
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Score on scale
Arm/Group | Arm A: Belantamab Mafodotin 2.5 Milligram (mg)/Kilogram (kg) Every 3 Weeks (Q3W) | Arm B: Belantamab Mafodotin 1.9 mg/kg Q3W | Arm C: Belantamab Mafodotin 2.5 mg/kg Every 6 Weeks (Q6W) | Arm D: Belantamab Mafodotin 1.9 mg/kg Q6W | Arm E: Belantamab Mafodotin 1.9 mg/kg Q6W (Based on OSDI + Visual Acuity [VA] Assessment)
Number analyzed (Participants) | 39 | 40 | 39 | 40 | 17
Score on scale | 3.68 (1.078) | 3.83 (1.017) | 3.87 (1.092) | 3.43 (1.031) | 3.64 (0.892)

9. Secondary Outcome: Duration of Corneal Events of Grade 2 or Above
Description: Duration of corneal events is defined for each participant as the sum of duration of all the corneal AEs. The duration is defined as time from onset of any corneal events (KVA scale) of Grade 2 or above to the first time resolution to baseline, Grade 1 or below. It required at least one day gap between the resolution of all events from first occurrence to the onset of next occurrence.
Time Frame: Up to 152 weeks
Population: as for outcome 7
Measure: Median (Full Range); unit: Days
Arm/Group | Arm A: Belantamab Mafodotin 2.5 Milligram (mg)/Kilogram (kg) Every 3 Weeks (Q3W) | Arm B: Belantamab Mafodotin 1.9 mg/kg Q3W | Arm C: Belantamab Mafodotin 2.5 mg/kg Every 6 Weeks (Q6W) | Arm D: Belantamab Mafodotin 1.9 mg/kg Q6W | Arm E: Belantamab Mafodotin 1.9 mg/kg Q6W (Based on OSDI + Visual Acuity [VA] Assessment)
Number analyzed (Participants) | 25 | 16 | 17 | 15 | 11
Days | 63.0 [22 to 296] | 67.5 [13 to 233] | 46.5 [20 to 162] | 53.5 [20 to 148] | 44.0 [21 to 274]

10. Secondary Outcome: Percentage of Time on Study With Grade 2 or Above Corneal Events
Description: It is defined as the percentage of time that a participant has corneal events out of the total time that a participant is on the study. Time with corneal events is defined as time from onset of any corneal events (KVA scale) of Grade 2 or above to the first-time resolution to baseline, Grade 1 or below.
Time Frame: Up to 152 weeks
Population: Safety Population. Only those participants who experienced corneal events of Grade 2 or above have been analyzed.
Measure: Median (Full Range); unit: Percentage of Time
Arm/Group | Arm A: Belantamab Mafodotin 2.5 Milligram (mg)/Kilogram (kg) Every 3 Weeks (Q3W) | Arm B: Belantamab Mafodotin 1.9 mg/kg Q3W | Arm C: Belantamab Mafodotin 2.5 mg/kg Every 6 Weeks (Q6W) | Arm D: Belantamab Mafodotin 1.9 mg/kg Q6W | Arm E: Belantamab Mafodotin 1.9 mg/kg Q6W (Based on OSDI + Visual Acuity [VA] Assessment)
Number analyzed (Participants) | 25 | 16 | 17 | 15 | 11
Percentage of Time | 23.27 [0.5 to 76.7] | 24.86 [5.1 to 69.1] | 18.99 [0.4 to 78.1] | 23.67 [5.5 to 85.6] | 35.63 [3.9 to 61.6]

11. Secondary Outcome: Number of Participants With Change in Best Corrected Visual Acuity Test (BCVA) Scores
Description: Change in BCVA is defined as change in logarithm of the minimum angle of resolution (logMAR) units compared with baseline or the first visit after the cataract surgery. BCVA score was calculated based on the Logarithm of the Minimum Angle of Resolution (logMAR score). Any change from baseline categories is presented for right and left eyes. No change/improved vision is defined as a change from baseline <0.1; a possible worsened vision is defined as a change from baseline >=0.1 to <=0.3; a definite worsened vision is defined as a change from baseline >0.3 logMAR score. Improvement in BCVA is represented by a reduction in logMAR score from baseline, while worsening in BCVA is represented by an increase in logMAR score from baseline.
Time Frame: Baseline (Day 1) and up to 152 weeks
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Belantamab Mafodotin 2.5 Milligram (mg)/Kilogram (kg) Every 3 Weeks (Q3W) | Arm B: Belantamab Mafodotin 1.9 mg/kg Q3W | Arm C: Belantamab Mafodotin 2.5 mg/kg Every 6 Weeks (Q6W) | Arm D: Belantamab Mafodotin 1.9 mg/kg Q6W | Arm E: Belantamab Mafodotin 1.9 mg/kg Q6W (Based on OSDI + Visual Acuity [VA] Assessment)
Number analyzed (Participants) | 22 | 24 | 23 | 29 | 11
Participants
  Left Eye: No change | 16 | 20 | 19 | 27 | 8
  Left Eye: Possible worsened vision | 2 | 3 | 3 | 1 | 1
  Left Eye: Definite worsened vision | 4 | 1 | 1 | 1 | 2
  Right Eye: number analyzed (Participants) | 21 | 24 | 23 | 29 | 11
  Right Eye: No change | 16 | 18 | 21 | 27 | 10
  Right Eye: Possible worsened vision | 4 | 5 | 2 | 2 | 1
  Right Eye: Definite worsened vision | 1 | 1 | 0 | 0 | 0

12. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants with a confirmed partial response (PR) or better (i.e., PR, very good partial response [VGPR], complete response [CR] and stringent complete response [sCR]), according to the International Myeloma Working Group (IMWG) Response Criteria. CR = negative immunofixation of serum and urine AND disappearance of any soft tissue plasmacytomas AND <5% plasmacytomas in the bone marrow; sCR=stringent complete response, CR as above PLUS normal serum free light-chain (FLC) assay ratio and absence of clonal cells in bone marrow by immunohistochemistry or immunofluorescence; VGPR = serum and urine M-component detectable by immunofixation but not on electrophoresis OR ≥ 90% reduction in serum M-component plus urine M-component <100 mg/24 h; PR = ≥50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by ≥90% or to <200 mg/24 h.
Time Frame: Up to 152 weeks
Population: Intent-to-Treat Population included all randomized participants, whether or not randomized treatment was administered.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Belantamab Mafodotin 2.5 Milligram (mg)/Kilogram (kg) Every 3 Weeks (Q3W) | Arm B: Belantamab Mafodotin 1.9 mg/kg Q3W | Arm C: Belantamab Mafodotin 2.5 mg/kg Every 6 Weeks (Q6W) | Arm D: Belantamab Mafodotin 1.9 mg/kg Q6W | Arm E: Belantamab Mafodotin 1.9 mg/kg Q6W (Based on OSDI + Visual Acuity [VA] Assessment)
Number analyzed (Participants) | 40 | 40 | 40 | 40 | 17
Percentage of participants | 33 [18.6 to 49.1] | 25 [12.7 to 41.2] | 28 [14.6 to 43.9] | 25 [12.7 to 41.2] | 18 [3.8 to 43.4]

13. Secondary Outcome: Percentage of Participants With a Confirmed VGPR or Better (i.e., VGPR, CR, and sCR)
Description: Percentage of participants with a confirmed VGPR or better defined as percentage of participant with confirmed VGPR, CR, and sCR, according to the 2016 IMWG response criteria. CR = negative immunofixation of serum and urine AND disappearance of any soft tissue plasmacytomas AND <5% plasmacytomas in the bone marrow; sCR=stringent complete response, CR as above PLUS normal serum free light-chain (FLC) assay ratio and absence of clonal cells in bone marrow by immunohistochemistry or immunofluorescence; VGPR = serum and urine M-component detectable by immunofixation but not on electrophoresis OR ≥ 90% reduction in serum M-component plus urine M-component <100 mg/24 h.
Time Frame: Up to 152 weeks
Population: Intent-to-Treat Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: Belantamab Mafodotin 2.5 Milligram (mg)/Kilogram (kg) Every 3 Weeks (Q3W) | Arm B: Belantamab Mafodotin 1.9 mg/kg Q3W | Arm C: Belantamab Mafodotin 2.5 mg/kg Every 6 Weeks (Q6W) | Arm D: Belantamab Mafodotin 1.9 mg/kg Q6W | Arm E: Belantamab Mafodotin 1.9 mg/kg Q6W (Based on OSDI + Visual Acuity [VA] Assessment)
Number analyzed (Participants) | 40 | 40 | 40 | 40 | 17
Percentage of participants | 25 [12.7 to 41.2] | 18 [7.3 to 32.8] | 8 [1.6 to 20.4] | 15 [5.7 to 29.8] | 18 [3.8 to 43.4]

14. Secondary Outcome: Time to Response (TTR)
Description: TTR defined as the time between the date of randomization and the first documented evidence of response (PR or better), among participants who achieve a response (i.e., confirmed PR or better), according to the 2016 IMWG response criteria. PR = ≥50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by ≥90% or to <200 mg/24 h.
Time Frame: Up to 152 weeks
Population: Intent-to-Treat Population. Only those participants with confirmed partial response (PR) or better (i.e., PR, VGPR, CR and sCR) have been analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Belantamab Mafodotin 2.5 Milligram (mg)/Kilogram (kg) Every 3 Weeks (Q3W) | Arm B: Belantamab Mafodotin 1.9 mg/kg Q3W | Arm C: Belantamab Mafodotin 2.5 mg/kg Every 6 Weeks (Q6W) | Arm D: Belantamab Mafodotin 1.9 mg/kg Q6W | Arm E: Belantamab Mafodotin 1.9 mg/kg Q6W (Based on OSDI + Visual Acuity [VA] Assessment)
Number analyzed (Participants) | 13 | 10 | 11 | 10 | 3
Months | 0.8 [0.7 to 1.4] | 1.1 [0.7 to 2.1] | 0.7 [0.7 to 0.9] | 0.8 [0.7 to 2.2] | 1.5 [0.8 to NA] — The upper limit of the 95% confidence interval was not estimable at the time of the final analysis due to an insufficient number of participants with events within the length of follow-up in assessing the number of events

15. Secondary Outcome: Duration of Response (DoR)
Description: DoR defined as the time from first documented evidence of PR or better until disease progression (PD) among responders according to the 2016 IMWG response criteria or death due to any cause. PR = ≥50% reduction of serum M-protein and reduction in 24-hour urinary M-protein by ≥90% or to <200 mg/24 h. PD= Increase of 25% from lowest confirmed response value in 1 or more of the following criteria: Serum M-protein with absolute increase of >= 0.5 g/dL; Serum M-protein increase >= 1 g/dL if the lowest M-component was >=5 g/dL; Urinary M-protein (absolute increase must be >= 200 mg per 24 h).
Time Frame: Up to 152 weeks
Population: Intent-to-Treat Population. Only those participants with confirmed PR or better (i.e., PR, VGPR, CR and sCR) have been analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Belantamab Mafodotin 2.5 Milligram (mg)/Kilogram (kg) Every 3 Weeks (Q3W) | Arm B: Belantamab Mafodotin 1.9 mg/kg Q3W | Arm C: Belantamab Mafodotin 2.5 mg/kg Every 6 Weeks (Q6W) | Arm D: Belantamab Mafodotin 1.9 mg/kg Q6W | Arm E: Belantamab Mafodotin 1.9 mg/kg Q6W (Based on OSDI + Visual Acuity [VA] Assessment)
Number analyzed (Participants) | 13 | 10 | 11 | 10 | 3
Months | 15.9 [4.9 to 21.4] | 22.1 [4.2 to NA] — The upper limit of 95% confidence interval was not estimable at the time of the final analysis due to an insufficient number of participants with events within the length of follow-up in assessing the number of events | 6.2 [2.1 to 20.7] | 7.8 [2.8 to 13.3] | 15.9 [NA to NA] — The lower and upper limit 95% confidence interval were not estimable at the time of the final analysis due to an insufficient number of participants with events within the length of follow-up in assessing the number of events

16. Secondary Outcome: Time to Progression (TTP)
Description: TTP defined as the time from randomization until the earliest date of documented PD or death due to PD, according to the 2016 IMWG response criteria. PD= Increase of 25% from lowest confirmed response value in 1 or more of the following criteria: Serum M-protein with absolute increase of >= 0.5 g/dL; Serum M-protein increase >= 1 g/dL if the lowest M-component was >=5 g/dL; Urinary M-protein (absolute increase must be >= 200 mg per 24 h).
Time Frame: Up to 152 weeks
Population: Intent-to-Treat Population. Only those participants with documented PD or death due to PD have been analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Belantamab Mafodotin 2.5 Milligram (mg)/Kilogram (kg) Every 3 Weeks (Q3W) | Arm B: Belantamab Mafodotin 1.9 mg/kg Q3W | Arm C: Belantamab Mafodotin 2.5 mg/kg Every 6 Weeks (Q6W) | Arm D: Belantamab Mafodotin 1.9 mg/kg Q6W | Arm E: Belantamab Mafodotin 1.9 mg/kg Q6W (Based on OSDI + Visual Acuity [VA] Assessment)
Number analyzed (Participants) | 26 | 29 | 28 | 32 | 10
Months | 6.0 [2.8 to 10.4] | 2.1 [1.0 to 9.1] | 2.8 [1.7 to 4.2] | 2.7 [1.9 to 5.6] | 2.9 [0.8 to 17.3]

17. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS defined as the time from randomization until the earliest date of documented PD, according to the 2016 IMWG response criteria, or death due to any cause. PD= Increase of 25% from lowest confirmed response value in 1 or more of the following criteria: Serum M-protein with absolute increase of >= 0.5 g/dL; Serum M-protein increase >= 1 g/dL if the lowest M-component was >=5 g/dL; Urinary M-protein (absolute increase must be >= 200 mg per 24 h).
Time Frame: Up to 152 weeks
Population: Intent-to-Treat Population. Only those participants with documented PD or death due to any cause have been analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Belantamab Mafodotin 2.5 Milligram (mg)/Kilogram (kg) Every 3 Weeks (Q3W) | Arm B: Belantamab Mafodotin 1.9 mg/kg Q3W | Arm C: Belantamab Mafodotin 2.5 mg/kg Every 6 Weeks (Q6W) | Arm D: Belantamab Mafodotin 1.9 mg/kg Q6W | Arm E: Belantamab Mafodotin 1.9 mg/kg Q6W (Based on OSDI + Visual Acuity [VA] Assessment)
Number analyzed (Participants) | 29 | 30 | 30 | 34 | 11
Months | 5.7 [2.8 to 9.0] | 2.1 [1.0 to 3.6] | 2.8 [1.4 to 3.5] | 2.7 [1.9 to 4.2] | 2.8 [0.8 to 17.3]

18. Secondary Outcome: Overall Survival (OS)
Description: OS defined as the time from randomization until the date of death due to any cause.
Time Frame: Up to 152 weeks
Population: Intent-to-Treat Population. Only those participants with documented death due to any cause have been analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Belantamab Mafodotin 2.5 Milligram (mg)/Kilogram (kg) Every 3 Weeks (Q3W) | Arm B: Belantamab Mafodotin 1.9 mg/kg Q3W | Arm C: Belantamab Mafodotin 2.5 mg/kg Every 6 Weeks (Q6W) | Arm D: Belantamab Mafodotin 1.9 mg/kg Q6W | Arm E: Belantamab Mafodotin 1.9 mg/kg Q6W (Based on OSDI + Visual Acuity [VA] Assessment)
Number analyzed (Participants) | 23 | 23 | 25 | 21 | 5
Months | 20.9 [8.1 to NA] — The upper limit of 95% confidence interval was not estimable at the time of the final analysis due to an insufficient number of participants with events within the length of follow-up in assessing the number of events. | 15.0 [7.6 to 20.1] | 13.5 [7.5 to 21.2] | 14.5 [7.7 to NA] — The upper limit of 95% confidence interval was not estimable at the time of the final analysis due to an insufficient number of participants with events within the length of follow-up in assessing the number of events. | NA [4.8 to NA] — The median and upper limit 95% confidence interval was not estimable at the time of the final analysis due to an insufficient number of participants with events within the length of follow-up in assessing the number of events.

19. Secondary Outcome: Percentage of Participants With AEs
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. AEs were coded using the standard Medical Dictionary for Regulatory Activities (MedDRA).
Time Frame: Up to 152 weeks
Population: Safety Population
Measure: Number; unit: Percentage of participants
Arm/Group | Arm A: Belantamab Mafodotin 2.5 Milligram (mg)/Kilogram (kg) Every 3 Weeks (Q3W) | Arm B: Belantamab Mafodotin 1.9 mg/kg Q3W | Arm C: Belantamab Mafodotin 2.5 mg/kg Every 6 Weeks (Q6W) | Arm D: Belantamab Mafodotin 1.9 mg/kg Q6W | Arm E: Belantamab Mafodotin 1.9 mg/kg Q6W (Based on OSDI + Visual Acuity [VA] Assessment)
Number analyzed (Participants) | 39 | 40 | 39 | 40 | 17
Percentage of participants | 100 | 100 | 100 | 100 | 100

20. Secondary Outcome: Percentage of Participants Requiring Dose Reduction, Dose Interruption/Delay, Permanent Treatment Discontinuation Due to Any AEs
Description: Percentage of participants requiring dose reduction, dose interruption/delay, permanent treatment discontinuation due to any AEs were presented. An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. AEs were coded using the standard MedDRA.
Time Frame: Up to 152 weeks
Population: Safety Population
Measure: Number; unit: Percentage of participants
Arm/Group | Arm A: Belantamab Mafodotin 2.5 Milligram (mg)/Kilogram (kg) Every 3 Weeks (Q3W) | Arm B: Belantamab Mafodotin 1.9 mg/kg Q3W | Arm C: Belantamab Mafodotin 2.5 mg/kg Every 6 Weeks (Q6W) | Arm D: Belantamab Mafodotin 1.9 mg/kg Q6W | Arm E: Belantamab Mafodotin 1.9 mg/kg Q6W (Based on OSDI + Visual Acuity [VA] Assessment)
Number analyzed (Participants) | 39 | 40 | 39 | 40 | 17
Percentage of participants
  Dose Reduction | 8 | 13 | 5 | 5 | 18
  Dose Interruption/Delay | 31 | 23 | 13 | 10 | 35
  Permanent Treatment Discontinuation | 10 | 8 | 10 | 5 | 18

21. Secondary Outcome: Number of Participants With Worst-Case Hematology Results by Maximum Grade Increase Post-Baseline Relative to Baseline
Description: Blood samples were collected for the analysis of hematology parameters. The parameters were graded according to CTCAE grades. Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe or medically significant but not immediately life-threatening; Grade 4: Life-threatening consequences; Grade 5: Death related to AE. Higher grades indicate greater severity and an increase in CTCAE grade was defined relative to the Baseline grade. Any worst-case post baseline increases in grade 1/2/3 to a grade of 4 are presented.
Time Frame: Up to 152 weeks
Population: Safety Population. Only those participants with data available for specified categories have been analyzed. Participants were counted more than once within some categories, so the percentages may not add to 100 percent (%).
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Belantamab Mafodotin 2.5 Milligram (mg)/Kilogram (kg) Every 3 Weeks (Q3W) | Arm B: Belantamab Mafodotin 1.9 mg/kg Q3W | Arm C: Belantamab Mafodotin 2.5 mg/kg Every 6 Weeks (Q6W) | Arm D: Belantamab Mafodotin 1.9 mg/kg Q6W | Arm E: Belantamab Mafodotin 1.9 mg/kg Q6W (Based on OSDI + Visual Acuity [VA] Assessment)
Number analyzed (Participants) | 38 | 39 | 38 | 40 | 16
Participants
  Eosinophilia, Increase to Grades 1 to 4: number analyzed (Participants) | 32 | 25 | 31 | 22 | 15
  Eosinophilia, Increase to Grades 1 to 4 | 3 | 1 | 2 | 1 | 0
  Eosinophilia, Increase to Grades 2 to 4: number analyzed (Participants) | 32 | 25 | 31 | 22 | 15
  Eosinophilia, Increase to Grades 2 to 4 | 0 | 0 | 0 | 0 | 0
  Eosinophilia, Increase to Grades 3 to 4: number analyzed (Participants) | 32 | 25 | 31 | 22 | 15
  Eosinophilia, Increase to Grades 3 to 4 | 0 | 0 | 0 | 0 | 0
  Anemia, Increase to Grades 1 to 4 | 17 | 15 | 20 | 15 | 6
  Anemia, Increase to Grades 2 to 4 | 16 | 14 | 17 | 14 | 5
  Anemia, Increase to Grades 3 to 4 | 10 | 9 | 11 | 9 | 4
  Hemoglobin increased, Increase to Grades 1 to 4 | 1 | 1 | 0 | 0 | 0
  Hemoglobin increased, Increase to Grades 2 to 4 | 0 | 0 | 0 | 0 | 0
  Hemoglobin increased, Increase to Grades 3 to 4 | 0 | 0 | 0 | 0 | 0
  Leukocytosis, Increase to Grades 1 to 4: number analyzed (Participants) | 38 | 39 | 37 | 40 | 16
  Leukocytosis, Increase to Grades 1 to 4 | 2 | 0 | 0 | 0 | 0
  Leukocytosis, Increase to Grades 2 to 4: number analyzed (Participants) | 38 | 39 | 37 | 40 | 16
  Leukocytosis, Increase to Grades 2 to 4 | 2 | 0 | 0 | 0 | 0
  Leukocytosis, Increase to Grades 3 to 4: number analyzed (Participants) | 38 | 39 | 37 | 40 | 16
  Leukocytosis, Increase to Grades 3 to 4 | 2 | 0 | 0 | 0 | 0
  White blood cell decreased, Increase to Grades 1 to 4: number analyzed (Participants) | 38 | 39 | 37 | 40 | 16
  White blood cell decreased, Increase to Grades 1 to 4 | 22 | 17 | 18 | 19 | 9
  White blood cell decreased, Increase to Grades 2 to 4: number analyzed (Participants) | 38 | 39 | 37 | 40 | 16
  White blood cell decreased, Increase to Grades 2 to 4 | 17 | 13 | 13 | 9 | 6
  White blood cell decreased, Increase to Grades 3 to 4: number analyzed (Participants) | 38 | 39 | 37 | 40 | 16
  White blood cell decreased, Increase to Grades 3 to 4 | 9 | 7 | 5 | 6 | 4
  Lymphocyte count decreased, Increase to Grades 1 to 4: number analyzed (Participants) | 33 | 28 | 32 | 28 | 15
  Lymphocyte count decreased, Increase to Grades 1 to 4 | 18 | 13 | 15 | 6 | 6
  Lymphocyte count decreased, Increase to Grades 2 to 4: number analyzed (Participants) | 33 | 28 | 32 | 28 | 15
  Lymphocyte count decreased, Increase to Grades 2 to 4 | 11 | 7 | 9 | 5 | 3
  Lymphocyte count decreased, Increase to Grades 3 to 4: number analyzed (Participants) | 33 | 28 | 32 | 28 | 15
  Lymphocyte count decreased, Increase to Grades 3 to 4 | 6 | 4 | 4 | 4 | 1
  Lymphocyte count increased, Increase to Grades 1 to 4: number analyzed (Participants) | 33 | 28 | 32 | 28 | 15
  Lymphocyte count increased, Increase to Grades 1 to 4 | 2 | 2 | 3 | 4 | 0
  Lymphocyte count increased, Increase to Grades 2 to 4: number analyzed (Participants) | 33 | 28 | 32 | 28 | 15
  Lymphocyte count increased, Increase to Grades 2 to 4 | 2 | 2 | 3 | 4 | 0
  Lymphocyte count increased, Increase to Grades 3 to 4: number analyzed (Participants) | 33 | 28 | 32 | 28 | 15
  Lymphocyte count increased, Increase to Grades 3 to 4 | 2 | 2 | 1 | 3 | 0
  Neutrophil count decreased, Increase to Grades 1 to 4: number analyzed (Participants) | 35 | 29 | 32 | 31 | 15
  Neutrophil count decreased, Increase to Grades 1 to 4 | 15 | 12 | 12 | 9 | 5
  Neutrophil count decreased, Increase to Grades 2 to 4: number analyzed (Participants) | 35 | 29 | 32 | 31 | 15
  Neutrophil count decreased, Increase to Grades 2 to 4 | 10 | 7 | 6 | 7 | 4
  Neutrophil count decreased, Increase to Grades 3 to 4: number analyzed (Participants) | 35 | 29 | 32 | 31 | 15
  Neutrophil count decreased, Increase to Grades 3 to 4 | 5 | 4 | 2 | 3 | 4
  Platelet count decreased, Increase to Grades 1 to 4: number analyzed (Participants) | 38 | 39 | 37 | 40 | 16
  Platelet count decreased, Increase to Grades 1 to 4 | 24 | 30 | 23 | 21 | 7
  Platelet count decreased, Increase to Grades 2 to 4: number analyzed (Participants) | 38 | 39 | 37 | 40 | 16
  Platelet count decreased, Increase to Grades 2 to 4 | 15 | 20 | 12 | 13 | 5
  Platelet count decreased, Increase to Grades 3 to 4: number analyzed (Participants) | 38 | 39 | 37 | 40 | 16
  Platelet count decreased, Increase to Grades 3 to 4 | 9 | 13 | 10 | 9 | 4

22. Secondary Outcome: Number of Participants With Worst-Case Clinical Chemistry Results by Maximum Grade Increase Post-Baseline Relative to Baseline
Description: Blood samples were collected for the analysis of clinical chemistry parameters. The parameters were graded according to CTCAE grades. Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe or medically significant but not immediately life-threatening; Grade 4: Life-threatening consequences; Grade 5: Death related to AE. Higher grades indicate greater severity and an increase in CTCAE grade was defined relative to the Baseline grade. Any worst-case post baseline increases in grade 1/2/3 to a grade of 4 are presented.
Time Frame: Up to 152 weeks
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Belantamab Mafodotin 2.5 Milligram (mg)/Kilogram (kg) Every 3 Weeks (Q3W) | Arm B: Belantamab Mafodotin 1.9 mg/kg Q3W | Arm C: Belantamab Mafodotin 2.5 mg/kg Every 6 Weeks (Q6W) | Arm D: Belantamab Mafodotin 1.9 mg/kg Q6W | Arm E: Belantamab Mafodotin 1.9 mg/kg Q6W (Based on OSDI + Visual Acuity [VA] Assessment)
Number analyzed (Participants) | 38 | 38 | 37 | 40 | 15
Participants
  Alanine aminotransferase increased, Increase to Grades 1 to 4: number analyzed (Participants) | 38 | 36 | 37 | 40 | 15
  Alanine aminotransferase increased, Increase to Grades 1 to 4 | 9 | 14 | 12 | 9 | 2
  Alanine aminotransferase increased, Increase to Grades 2 to 4: number analyzed (Participants) | 38 | 36 | 37 | 40 | 15
  Alanine aminotransferase increased, Increase to Grades 2 to 4 | 2 | 3 | 1 | 1 | 0
  Alanine aminotransferase increased, Increase to Grades 3 to 4: number analyzed (Participants) | 38 | 36 | 37 | 40 | 15
  Alanine aminotransferase increased, Increase to Grades 3 to 4 | 1 | 0 | 1 | 0 | 0
  Hypoalbuminemia, Increase to Grades 1 to 4: number analyzed (Participants) | 38 | 38 | 36 | 39 | 15
  Hypoalbuminemia, Increase to Grades 1 to 4 | 19 | 15 | 14 | 13 | 7
  Hypoalbuminemia, Increase to Grades 2 to 4: number analyzed (Participants) | 38 | 38 | 36 | 39 | 15
  Hypoalbuminemia, Increase to Grades 2 to 4 | 6 | 9 | 11 | 6 | 2
  Hypoalbuminemia, Increase to Grades 3 to 4: number analyzed (Participants) | 38 | 38 | 36 | 39 | 15
  Hypoalbuminemia, Increase to Grades 3 to 4 | 1 | 2 | 1 | 1 | 0
  Alkaline phosphatase increased, Increase to Grades 1 to 4: number analyzed (Participants) | 38 | 36 | 35 | 40 | 15
  Alkaline phosphatase increased, Increase to Grades 1 to 4 | 10 | 15 | 8 | 9 | 3
  Alkaline phosphatase increased, Increase to Grades 2 to 4: number analyzed (Participants) | 38 | 36 | 35 | 40 | 15
  Alkaline phosphatase increased, Increase to Grades 2 to 4 | 1 | 2 | 1 | 1 | 0
  Alkaline phosphatase increased, Increase to Grades 3 to 4: number analyzed (Participants) | 38 | 36 | 35 | 40 | 15
  Alkaline phosphatase increased, Increase to Grades 3 to 4 | 0 | 0 | 0 | 1 | 0
  Aspartate aminotransferase increased, Increase to Grades 1 to 4: number analyzed (Participants) | 38 | 36 | 36 | 40 | 15
  Aspartate aminotransferase increased, Increase to Grades 1 to 4 | 20 | 23 | 22 | 14 | 3
  Aspartate aminotransferase increased, Increase to Grades 2 to 4: number analyzed (Participants) | 38 | 36 | 36 | 40 | 15
  Aspartate aminotransferase increased, Increase to Grades 2 to 4 | 4 | 3 | 2 | 1 | 0
  Aspartate aminotransferase increased, Increase to Grades 3 to 4: number analyzed (Participants) | 38 | 36 | 36 | 40 | 15
  Aspartate aminotransferase increased, Increase to Grades 3 to 4 | 1 | 0 | 1 | 0 | 0
  Blood bilirubin increased, Increase to Grades 1 to 4: number analyzed (Participants) | 38 | 37 | 36 | 40 | 15
  Blood bilirubin increased, Increase to Grades 1 to 4 | 4 | 4 | 4 | 3 | 3
  Blood bilirubin increased, Increase to Grades 2 to 4: number analyzed (Participants) | 38 | 37 | 36 | 40 | 15
  Blood bilirubin increased, Increase to Grades 2 to 4 | 2 | 0 | 0 | 0 | 1
  Blood bilirubin increased, Increase to Grades 3 to 4: number analyzed (Participants) | 38 | 37 | 36 | 40 | 15
  Blood bilirubin increased, Increase to Grades 3 to 4 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia, Increase to Grades 1 to 4: number analyzed (Participants) | 38 | 38 | 36 | 39 | 15
  Hypercalcemia, Increase to Grades 1 to 4 | 14 | 13 | 15 | 12 | 4
  Hypercalcemia, Increase to Grades 2 to 4: number analyzed (Participants) | 38 | 38 | 36 | 39 | 15
  Hypercalcemia, Increase to Grades 2 to 4 | 3 | 2 | 5 | 3 | 1
  Hypercalcemia, Increase to Grades 3 to 4: number analyzed (Participants) | 38 | 38 | 36 | 39 | 15
  Hypercalcemia, Increase to Grades 3 to 4 | 3 | 1 | 2 | 2 | 1
  Hypocalcemia, Increase to Grades 1 to 4: number analyzed (Participants) | 38 | 38 | 36 | 39 | 15
  Hypocalcemia, Increase to Grades 1 to 4 | 12 | 16 | 8 | 10 | 6
  Hypocalcemia, Increase to Grades 2 to 4: number analyzed (Participants) | 38 | 38 | 36 | 39 | 15
  Hypocalcemia, Increase to Grades 2 to 4 | 3 | 4 | 3 | 2 | 1
  Hypocalcemia, Increase to Grades 3 to 4: number analyzed (Participants) | 38 | 38 | 36 | 39 | 15
  Hypocalcemia, Increase to Grades 3 to 4 | 1 | 3 | 1 | 1 | 0
  CPK increased, Increase to Grades 1 to 4: number analyzed (Participants) | 38 | 36 | 32 | 38 | 15
  CPK increased, Increase to Grades 1 to 4 | 11 | 8 | 5 | 6 | 2
  CPK increased, Increase to Grades 2 to 4: number analyzed (Participants) | 38 | 36 | 32 | 38 | 15
  CPK increased, Increase to Grades 2 to 4 | 5 | 3 | 1 | 0 | 0
  CPK increased, Increase to Grades 3 to 4: number analyzed (Participants) | 38 | 36 | 32 | 38 | 15
  CPK increased, Increase to Grades 3 to 4 | 2 | 1 | 0 | 0 | 0
  Creatinine increased, Increase to Grades 1 to 4 | 14 | 18 | 18 | 15 | 7
  Creatinine increased, Increase to Grades 2 to 4 | 6 | 9 | 6 | 7 | 2
  Creatinine increased, Increase to Grades 3 to 4 | 0 | 0 | 1 | 0 | 1
  Chronic Kidney Disease, Increase to Grades 1 to 4: number analyzed (Participants) | 19 | 20 | 21 | 23 | 9
  Chronic Kidney Disease, Increase to Grades 1 to 4 | 6 | 8 | 8 | 8 | 4
  Chronic Kidney Disease, Increase to Grades 2 to 4: number analyzed (Participants) | 19 | 20 | 21 | 23 | 9
  Chronic Kidney Disease, Increase to Grades 2 to 4 | 6 | 6 | 8 | 8 | 4
  Chronic Kidney Disease, Increase to Grades 3 to 4: number analyzed (Participants) | 19 | 20 | 21 | 23 | 9
  Chronic Kidney Disease, Increase to Grades 3 to 4 | 3 | 3 | 1 | 3 | 2
  GGT increased, Increase to Grades 1 to 4: number analyzed (Participants) | 38 | 36 | 36 | 40 | 13
  GGT increased, Increase to Grades 1 to 4 | 17 | 16 | 16 | 9 | 5
  GGT increased, Increase to Grades 2 to 4: number analyzed (Participants) | 38 | 36 | 36 | 40 | 13
  GGT increased, Increase to Grades 2 to 4 | 10 | 7 | 3 | 7 | 1
  GGT increased, Increase to Grades 3 to 4: number analyzed (Participants) | 38 | 36 | 36 | 40 | 13
  GGT increased, Increase to Grades 3 to 4 | 2 | 3 | 1 | 3 | 0
  Blood lactate dehydrogenase increased, Increase to Grades 1 to 4: number analyzed (Participants) | 38 | 37 | 36 | 40 | 15
  Blood lactate dehydrogenase increased, Increase to Grades 1 to 4 | 20 | 19 | 19 | 15 | 6
  Blood lactate dehydrogenase increased, Increase to Grades 2 to 4: number analyzed (Participants) | 38 | 37 | 36 | 40 | 15
  Blood lactate dehydrogenase increased, Increase to Grades 2 to 4 | 0 | 0 | 0 | 0 | 0
  Blood lactate dehydrogenase increased, Increase to Grades 3 to 4: number analyzed (Participants) | 38 | 37 | 36 | 40 | 15
  Blood lactate dehydrogenase increased, Increase to Grades 3 to 4 | 0 | 0 | 0 | 0 | 0
  Hypermagnesemia, Increase to Grades 1 to 4: number analyzed (Participants) | 38 | 36 | 35 | 39 | 15
  Hypermagnesemia, Increase to Grades 1 to 4 | 2 | 3 | 3 | 2 | 0
  Hypermagnesemia, Increase to Grades 2 to 4: number analyzed (Participants) | 38 | 36 | 35 | 39 | 15
  Hypermagnesemia, Increase to Grades 2 to 4 | 0 | 2 | 2 | 1 | 0
  Hypermagnesemia, Increase to Grades 3 to 4: number analyzed (Participants) | 38 | 36 | 35 | 39 | 15
  Hypermagnesemia, Increase to Grades 3 to 4 | 0 | 2 | 2 | 1 | 0
  Hypomagnesemia, Increase to Grades 1 to 4: number analyzed (Participants) | 38 | 36 | 35 | 39 | 15
  Hypomagnesemia, Increase to Grades 1 to 4 | 7 | 3 | 5 | 8 | 2
  Hypomagnesemia, Increase to Grades 2 to 4: number analyzed (Participants) | 38 | 36 | 35 | 39 | 15
  Hypomagnesemia, Increase to Grades 2 to 4 | 1 | 0 | 0 | 1 | 0
  Hypomagnesemia, Increase to Grades 3 to 4: number analyzed (Participants) | 38 | 36 | 35 | 39 | 15
  Hypomagnesemia, Increase to Grades 3 to 4 | 1 | 0 | 0 | 0 | 0
  Hyperkalemia, Increase to Grades 1 to 4: number analyzed (Participants) | 38 | 37 | 37 | 40 | 15
  Hyperkalemia, Increase to Grades 1 to 4 | 4 | 6 | 7 | 1 | 2
  Hyperkalemia, Increase to Grades 2 to 4: number analyzed (Participants) | 38 | 37 | 37 | 40 | 15
  Hyperkalemia, Increase to Grades 2 to 4 | 1 | 2 | 2 | 0 | 0
  Hyperkalemia, Increase to Grades 3 to 4: number analyzed (Participants) | 38 | 37 | 37 | 40 | 15
  Hyperkalemia, Increase to Grades 3 to 4 | 1 | 1 | 1 | 0 | 0
  Hypernatremia, Increase to Grades 1 to 4 | 4 | 4 | 3 | 5 | 3
  Hypernatremia, Increase to Grades 2 to 4 | 1 | 2 | 0 | 1 | 1
  Hypernatremia, Increase to Grades 3 to 4 | 1 | 2 | 0 | 1 | 1

23. Secondary Outcome: Number of Participants With Post-baseline Positive Anti-drug Antibodies (ADAs) Against Belantamab Mafodotin
Description: Serum samples collected for the analysis of the presence of ADAs using validated immunoassays. All samples were tested in screening assay, and positive samples were further characterized for antibody titers. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits.
Time Frame: Baseline (Day 1) and up to 152 weeks
Population: Safety Population. Only those participants with data available at specified time points have been analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Belantamab Mafodotin 2.5 Milligram (mg)/Kilogram (kg) Every 3 Weeks (Q3W) | Arm B: Belantamab Mafodotin 1.9 mg/kg Q3W | Arm C: Belantamab Mafodotin 2.5 mg/kg Every 6 Weeks (Q6W) | Arm D: Belantamab Mafodotin 1.9 mg/kg Q6W | Arm E: Belantamab Mafodotin 1.9 mg/kg Q6W (Based on OSDI + Visual Acuity [VA] Assessment)
Number analyzed (Participants) | 37 | 37 | 32 | 36 | 15
Participants | 0 | 0 | 0 | 0 | 0

24. Secondary Outcome: Titers of ADAs Against Belantamab Mafodotin
Description: Serum samples collected for the analysis of the presence of ADAs using validated immunoassays. All samples were to be further tested in screening assay, and positive samples were further to be characterized for antibody titers.
Time Frame: Up to 152 weeks
Population: Safety Population. There were no participants with positive ADA results. Hence the titer (concentration) of ADA was not collected.
Arm/Group | Arm A: Belantamab Mafodotin 2.5 Milligram (mg)/Kilogram (kg) Every 3 Weeks (Q3W) | Arm B: Belantamab Mafodotin 1.9 mg/kg Q3W | Arm C: Belantamab Mafodotin 2.5 mg/kg Every 6 Weeks (Q6W) | Arm D: Belantamab Mafodotin 1.9 mg/kg Q6W | Arm E: Belantamab Mafodotin 1.9 mg/kg Q6W (Based on OSDI + Visual Acuity [VA] Assessment)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

25. Secondary Outcome: Maximum Observed Concentration (Cmax) for Belantamab Mafodotin Antibody-drug Conjugate (ADC)
Description: Plasma samples were collected for PK analysis for belantamab mafodotin antibody-drug conjugate (ADC).
Time Frame: Cycle(C)1 Day(D) 1 Pre-dose, End of Infusion (EOI), Start of Infusion (SOI) + 2 hours (H); C1D2 SOI+24H; C1D4; C1D8-15
Population: Pharmacokinetic (PK) Population included all participants in the Safety Population from whom at least 1 post-treatment PK sample was obtained and analyzed. One Participant was randomized in Arm A but inadvertently given Arm B treatment at Cycle 1. Hence included in Arm B for PK analyses.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram/ millilitre (ug/mL)
Arm/Group | Arm A: Belantamab Mafodotin 2.5 Milligram (mg)/Kilogram (kg) Every 3 Weeks (Q3W) | Arm B: Belantamab Mafodotin 1.9 mg/kg Q3W | Arm C: Belantamab Mafodotin 2.5 mg/kg Every 6 Weeks (Q6W) | Arm D: Belantamab Mafodotin 1.9 mg/kg Q6W | Arm E: Belantamab Mafodotin 1.9 mg/kg Q6W (Based on OSDI + Visual Acuity [VA] Assessment)
Number analyzed (Participants) | 38 | 41 | 39 | 40 | 17
Microgram/ millilitre (ug/mL) | 44.8 (22.8) | 33.1 (23.2) | 42.1 (24.7) | 33.1 (18.3) | 34.1 (26.8)

26. Secondary Outcome: Concentration at 21 Days for Belantamab Mafodotin ADC
Description: Plasma samples were collected for PK analysis for belantamab mafodotin ADC.
Time Frame: At 21 days
Population: Pharmacokinetic (PK) Population. One Participant was randomized in Arm A but inadvertently given Arm B treatment at Cycle 1. Hence included in Arm B for PK analyses.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Arm A: Belantamab Mafodotin 2.5 Milligram (mg)/Kilogram (kg) Every 3 Weeks (Q3W) | Arm B: Belantamab Mafodotin 1.9 mg/kg Q3W | Arm C: Belantamab Mafodotin 2.5 mg/kg Every 6 Weeks (Q6W) | Arm D: Belantamab Mafodotin 1.9 mg/kg Q6W | Arm E: Belantamab Mafodotin 1.9 mg/kg Q6W (Based on OSDI + Visual Acuity [VA] Assessment)
Number analyzed (Participants) | 38 | 41 | 39 | 40 | 17
ug/mL | 2.28 (56.7) | 1.5 (62.4) | 1.94 (69.3) | 1.69 (50.2) | 1.53 (62.1)

27. Secondary Outcome: Average Concentration Over 21 Days (Cavg) for Belantamab Mafodotin ADC
Description: Plasma samples were collected for PK analysis for belantamab mafodotin ADC.
Time Frame: C1 D1 Pre-dose, EOI, SOI + 2H; C1D2 SOI+24H; C1D4; C1D8-15, D21
Population: as for outcome 26
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Arm A: Belantamab Mafodotin 2.5 Milligram (mg)/Kilogram (kg) Every 3 Weeks (Q3W) | Arm B: Belantamab Mafodotin 1.9 mg/kg Q3W | Arm C: Belantamab Mafodotin 2.5 mg/kg Every 6 Weeks (Q6W) | Arm D: Belantamab Mafodotin 1.9 mg/kg Q6W | Arm E: Belantamab Mafodotin 1.9 mg/kg Q6W (Based on OSDI + Visual Acuity [VA] Assessment)
Number analyzed (Participants) | 38 | 41 | 39 | 40 | 17
ug/mL | 8.4 (32.2) | 5.98 (34.6) | 7.71 (38.6) | 6.3 (27.1) | 6.11 (40.6)

28. Secondary Outcome: Area Under the Concentration-time Curve (AUC) (0-504h) of Belantamab Mafodotin ADC
Description: Plasma samples were collected to determine the area under the concentration-time curve (AUC) (0-504h) of Belantamab mafodotin ADC.
Time Frame: C1 D1 Pre-dose, EOI, SOI + 2H; C1D2 SOI+24H; C1D4; C1D8-15, D21
Population: as for outcome 26
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms* hour/ millilitre (ug*h/mL)
Arm/Group | Arm A: Belantamab Mafodotin 2.5 Milligram (mg)/Kilogram (kg) Every 3 Weeks (Q3W) | Arm B: Belantamab Mafodotin 1.9 mg/kg Q3W | Arm C: Belantamab Mafodotin 2.5 mg/kg Every 6 Weeks (Q6W) | Arm D: Belantamab Mafodotin 1.9 mg/kg Q6W | Arm E: Belantamab Mafodotin 1.9 mg/kg Q6W (Based on OSDI + Visual Acuity [VA] Assessment)
Number analyzed (Participants) | 38 | 41 | 39 | 40 | 17
micrograms* hour/ millilitre (ug*h/mL) | 4233 (32.2) | 3013 (34.6) | 3886 (38.6) | 3173 (27.1) | 3079 (40.6)

29. Secondary Outcome: Half-life (t1/2) of Belantamab Mafodotin ADC
Description: Plasma samples were collected for PK analysis of Belantamab mafodotin ADC
Time Frame: C1 D1 Pre-dose, EOI, SOI + 2H; C1D2 SOI+24H; C1D4; C1D8-15
Population: as for outcome 26
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Days
Arm/Group | Arm A: Belantamab Mafodotin 2.5 Milligram (mg)/Kilogram (kg) Every 3 Weeks (Q3W) | Arm B: Belantamab Mafodotin 1.9 mg/kg Q3W | Arm C: Belantamab Mafodotin 2.5 mg/kg Every 6 Weeks (Q6W) | Arm D: Belantamab Mafodotin 1.9 mg/kg Q6W | Arm E: Belantamab Mafodotin 1.9 mg/kg Q6W (Based on OSDI + Visual Acuity [VA] Assessment)
Number analyzed (Participants) | 38 | 41 | 39 | 40 | 17
Days | 13 (30.5) | 12 (32.1) | 12 (40) | 12 (34.2) | 13 (41.3)

30. Secondary Outcome: Clearance (CL) for Belantamab Mafodotin ADC
Description: Plasma samples were collected for PK analysis for belantamab mafodotin ADC.
Time Frame: C1 D1 Pre-dose, EOI, SOI + 2H; C1D2 SOI+24H; C1D4; C1D8-15
Population: as for outcome 26
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter/ days
Arm/Group | Arm A: Belantamab Mafodotin 2.5 Milligram (mg)/Kilogram (kg) Every 3 Weeks (Q3W) | Arm B: Belantamab Mafodotin 1.9 mg/kg Q3W | Arm C: Belantamab Mafodotin 2.5 mg/kg Every 6 Weeks (Q6W) | Arm D: Belantamab Mafodotin 1.9 mg/kg Q6W | Arm E: Belantamab Mafodotin 1.9 mg/kg Q6W (Based on OSDI + Visual Acuity [VA] Assessment)
Number analyzed (Participants) | 38 | 41 | 39 | 40 | 17
Liter/ days | 0.8 (38.3) | 0.83 (57.1) | 0.84 (47.7) | 0.74 (53.3) | 0.86 (59.7)

31. Secondary Outcome: Steady-state Volume of Distribution (Vss) for Belantamab Mafodotin ADC
Description: Plasma samples were collected for PK analysis for belantamab mafodotin ADC.
Time Frame: C1 D1 Pre-dose, EOI, SOI + 2H; C1D2 SOI+24H; C1D4; C1D8-15
Population: as for outcome 26
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Arm A: Belantamab Mafodotin 2.5 Milligram (mg)/Kilogram (kg) Every 3 Weeks (Q3W) | Arm B: Belantamab Mafodotin 1.9 mg/kg Q3W | Arm C: Belantamab Mafodotin 2.5 mg/kg Every 6 Weeks (Q6W) | Arm D: Belantamab Mafodotin 1.9 mg/kg Q6W | Arm E: Belantamab Mafodotin 1.9 mg/kg Q6W (Based on OSDI + Visual Acuity [VA] Assessment)
Number analyzed (Participants) | 38 | 41 | 39 | 40 | 17
Liter | 10.0 (19.6) | 9.3 (26.4) | 9.4 (26.9) | 8.9 (25.4) | 10.0 (16.1)

ADVERSE EVENTS:
Time Frame: All-cause mortality, Serious adverse events (SAEs) and non-serious AEs (Non SAEs) were collected up to 152 weeks.
Description: All-cause mortality was collected based on ITT Population included all randomized participants, whether or not randomized treatment was administered. SAEs and non-SAEs were collected based on Safety Population included all randomized participants who received at least 1 dose of study treatment. The results presented are based on data cut-off date 30 Jan 2025 and additional safety results will be updated within a year of study completion.
Arm/Group | Arm A: Belantamab Mafodotin 2.5 Milligram (mg)/Kilogram (kg) Every 3 Weeks (Q3W) | Arm B: Belantamab Mafodotin 1.9 mg/kg Q3W | Arm C: Belantamab Mafodotin 2.5 mg/kg Every 6 Weeks (Q6W) | Arm D: Belantamab Mafodotin 1.9 mg/kg Q6W | Arm E: Belantamab Mafodotin 1.9 mg/kg Q6W (Based on OSDI + Visual Acuity [VA] Assessment)
All-Cause Mortality (participants affected / at risk) | 23/40 | 23/40 | 25/40 | 21/40 | 5/17
Serious Adverse Events (participants affected / at risk) | 17/39 | 17/40 | 21/39 | 16/40 | 4/17
Other Adverse Events (participants affected / at risk) | 38/39 | 36/40 | 36/39 | 40/40 | 16/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Belantamab Mafodotin 2.5 Milligram (mg)/Kilogram (kg) Every 3 Weeks (Q3W) (N=39) | Arm B: Belantamab Mafodotin 1.9 mg/kg Q3W (N=40) | Arm C: Belantamab Mafodotin 2.5 mg/kg Every 6 Weeks (Q6W) (N=39) | Arm D: Belantamab Mafodotin 1.9 mg/kg Q6W (N=40) | Arm E: Belantamab Mafodotin 1.9 mg/kg Q6W (Based on OSDI + Visual Acuity [VA] Assessment) (N=17)
Pneumonia (Infections and infestations) | 2 (2) | 3 (5) | 3 (3) | 2 (2) | 1 (2)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Streptococcal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronavirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatitis B reactivation (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Metapneumovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia cytomegaloviral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia parainfluenzae viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Vascular device infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 4 (4) | 2 (2) | 2 (2) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Anaemia macrocytic (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
General physical health deterioration (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Disease progression (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Organ failure (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Systemic inflammatory response syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infected neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bone lesion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic venous thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Belantamab Mafodotin 2.5 Milligram (mg)/Kilogram (kg) Every 3 Weeks (Q3W) (N=39) | Arm B: Belantamab Mafodotin 1.9 mg/kg Q3W (N=40) | Arm C: Belantamab Mafodotin 2.5 mg/kg Every 6 Weeks (Q6W) (N=39) | Arm D: Belantamab Mafodotin 1.9 mg/kg Q6W (N=40) | Arm E: Belantamab Mafodotin 1.9 mg/kg Q6W (Based on OSDI + Visual Acuity [VA] Assessment) (N=17)
Anaemia (Blood and lymphatic system disorders) | 9 (16) | 12 (15) | 12 (13) | 15 (23) | 4 (4)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 8 (11) | 3 (3) | 7 (8) | 4 (4)
Thrombocytopenia (Blood and lymphatic system disorders) | 11 (17) | 17 (26) | 13 (20) | 10 (14) | 4 (4)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 5 (7) | 4 (4) | 2 (3) | 7 (9) | 3 (3)
Corneal epithelial microcysts (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Corneal erosion (Eye disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 15 (25) | 12 (17) | 12 (33) | 12 (17) | 8 (14)
Eye irritation (Eye disorders) | 11 (20) | 9 (19) | 11 (32) | 11 (21) | 5 (11)
Eye pain (Eye disorders) | 9 (13) | 2 (3) | 6 (25) | 4 (4) | 3 (3)
Eye pruritus (Eye disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eyelid irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Foreign body sensation in eyes (Eye disorders) | 7 (12) | 7 (14) | 11 (35) | 5 (8) | 3 (10)
Lacrimation increased (Eye disorders) | 3 (4) | 4 (4) | 0 (0) | 2 (3) | 0 (0)
Photophobia (Eye disorders) | 8 (12) | 10 (19) | 10 (19) | 3 (3) | 5 (12)
Punctate keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Trichiasis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ulcerative keratitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Vision blurred (Eye disorders) | 16 (36) | 12 (33) | 18 (53) | 11 (19) | 9 (22)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 6 (7) | 2 (2) | 6 (6) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 2 (3) | 4 (4) | 4 (4) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (4) | 3 (4) | 8 (9) | 3 (3) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 1 (1)
Asthenia (General disorders) | 2 (2) | 3 (3) | 3 (3) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Fatigue (General disorders) | 6 (6) | 6 (6) | 4 (5) | 1 (2) | 1 (1)
Pyrexia (General disorders) | 4 (4) | 3 (3) | 7 (7) | 3 (3) | 2 (2)
Sensation of foreign body (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Swelling (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 5 (5) | 1 (1) | 2 (2) | 3 (3) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (2)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Periorbital cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 3 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 8 (9) | 4 (5) | 3 (3) | 2 (2) | 1 (1)
Urinary tract infection (Infections and infestations) | 6 (6) | 3 (3) | 1 (1) | 1 (1) | 0 (0)
Eye injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 5 (6) | 2 (3) | 2 (3) | 5 (5) | 2 (2)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (3) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 4 (6) | 6 (8) | 4 (5) | 5 (6) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 2 (3) | 1 (3) | 2 (2) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 2 (8) | 0 (0) | 2 (2) | 0 (0)
Blood creatinine increased (Investigations) | 1 (2) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 6 (6) | 3 (8) | 3 (3) | 2 (2) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 3 (3) | 4 (4) | 3 (3) | 2 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (5) | 5 (7) | 2 (2) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (4) | 4 (5) | 4 (4) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4) | 3 (3) | 5 (5) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 5 (5) | 2 (3) | 2 (2) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Ocular neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1) | 3 (3) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Intensive care unit delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 2 (3) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 2 (2) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 3 (3) | 1 (1) | 3 (3) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2024-06-25): https://cdn.clinicaltrials.gov/large-docs/58/NCT05064358/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-18): https://cdn.clinicaltrials.gov/large-docs/58/NCT05064358/SAP_001.pdf